CLINICAL TRIAL: NCT00533208
Title: MK0524 Seasonal Allergic Rhinitis Study (0524-005)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524-005; 2007_616
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Seasonal Allergies
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — MK-0524

INTERVENTIONS:
Drug: MK0524

SUMMARY:
To assess the efficacy of MK0524 on seasonal allergies.

ELIGIBILITY:
Inclusion Criteria:

* Person has had at least 2 years of seasonal allergies
* Person has had a positive skin test to at least 1 of the allergens of the season
* Person is a non-smoker

Exclusion Criteria:

* Person has been hospitalized within the last 4 weeks
* Person is a female who has had a baby within the last 8 weeks or is still breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Actual)
Dates: Start 2003-07; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Philip G, van Adelsberg J, Loeys T, Liu N, Wong P, Lai E, Dass SB, Reiss TF. Clinical studies of the DP1 antagonist laropiprant in asthma and allergic rhinitis. J Allergy Clin Immunol. 2009 Nov;124(5):942-8.e1-9. doi: 10.1016/j.jaci.2009.07.006. Epub 2009 Sep 12. PMID 19748656